CLINICAL TRIAL: NCT01201148
Title: A Study of Transcranial Electrical Stimulation (TES) for the Treatment of Depression
Brief Title: Open Pilot Trial of TES for Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10231
Record Dates: First submitted 2010-09-08; First posted 2010-09-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Major Depression
Keywords: depression; transcranial direct current stimulation (tDCS); random noise stimulation; oscillatory tDCS; intermittent tDCS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oscillating or intermittent tDCS (Experimental)
  Interventions: Device: tDCS (Eldith DC-Stimulator (CE certified))

INTERVENTIONS:
Device: tDCS (Eldith DC-Stimulator (CE certified)) — For participants receiving intermittent tDCS or oscillating TES, one electrode will be placed over the left pF3 electrode site (overlying the left dorsolateral prefrontal cortex and identified on the scalp using an EEG cap based on the 10/20 system) and the other over the right temporal area.

SUMMARY:
This study will investigate whether using oscillating TES (random noise stimulation) or intermittent tDCS will have greater antidepressant effects in depressed subjects, compared to standard tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets criteria for a DSM-IV Major Depressive episode.

Exclusion Criteria:

* Diagnosis (as defined by DSM-IV) of: any psychotic disorder (lifetime); bipolar disorder; eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder (current or within the past year); mental retardation.
* Subject has not responded adequately to standard tDCS or is not appropriate for trial of standard tDCS (eg depression too chronic in duration)
* Total MADRS depression score of 20 or more
* History of drug or alcohol abuse or dependence (as per DSM-IV criteria) within the last 3 months (except nicotine and caffeine).
* Inadequate response to ECT in the current episode of depression.
* Subject is on regular benzodiazepine medication which it is not clinically appropriate to discontinue.
* Subject requires a rapid clinical response due to inanition, psychosis or high suicide risk.
* Neurological disorder or insult, e.g., recent stroke (CVA), which places subject at risk of seizure or neuronal damage with TES.
* Subject has metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
* Female subject who is pregnant. However, women of child bearing age are eligible if they have the pregnancy test but will be excluded if they are sexually active and not using reliable contraception (urine test for pregnancy will be used if appropriate).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, Principal Investigator — School of Psychiatry, University of New South Wales
Locations (1):
- Black Dog Institute, Sydney, New South Wales, Australia